CLINICAL TRIAL: NCT03147950
Title: Prone Versus Prone-Flexed Position For Percutaneous Nephrolithotomy (PCNL) Comparing Efficacy and Complication According to Clavien-Dindo Classification Score Randomised Controlled Study
Brief Title: Prone Versus Prone-Flexed Position For Percutaneous Nephrolithotomy (PCNL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F-Prone PNL
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Percutaneous Nephrolithotomy (PCNL); Prone Position; Prone-Flexed Position; Complication of Surgical Procedure
Keywords: Prone-Flexed Position; Percutaneous Nephrolithotomy (PCNL); Clavien-Dindo Classification Score

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone-Flexed PCNL (Active Comparator): Prone-Flexed Position For Percutaneous Nephrolithotomy (PCNL)
  Interventions: Procedure: Prone-Flexed PCNL
- Prone PCNL (Active Comparator): Prone Position For Percutaneous Nephrolithotomy (PCNL)
  Interventions: Procedure: Prone PCNL

INTERVENTIONS:
Procedure: Prone-Flexed PCNL — Prone-Flexed Position For Percutaneous Nephrolithotomy (PCNL)
  Other Names: Prone-Flexed Percutaneous Nephrolithotomy
  Arms: Prone-Flexed PCNL
Procedure: Prone PCNL — Prone Position For Percutaneous Nephrolithotomy (PCNL)
  Other Names: Prone Percutaneous Nephrolithotomy
  Arms: Prone PCNL

SUMMARY:
compare the prone with the prone-flexed position accessibility of upper and middle calyceal approach by subcostal puncture and PCNL reporting complications using the Clavien-Dindo system with Categorisation of PCNL-specific complications according to Clavien-Dindo classification score

ELIGIBILITY:
Inclusion Criteria:

* Large renal pelvic stone
* Upper calyceal stone
* Middle calyceal stone

Exclusion Criteria:

* lower calyceal stone
* Bilateral simultaneous PCNL
* Need for 3 percutaneous tracts intraoperative
* Morbid obesity (BMI >40)
* Non opaque renal stones.
* Refuse to complete study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the prone with the prone-flexed position for PCNL reporting complications | 1 year
  Outcome measures by using the clavien dindo classification system

SECONDARY OUTCOMES:
Assessment of stone free rate (SFR) of the two groups | 1 year
  Outcome measures by stone fragment residual ≤ 2 mm by computed tomography (CT)
Asses the easiness of accessibility of the targeted stone | 1 year
  Outcome measures by counting number and site of puncture trial

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shoma, MD, Study Chair — Urology and Nephrology center; Ahmed Elassmy, MD, Study Director — Urology and Nephrology center; Nasr Eltabey, MD, Study Director — Urology and Nephrology center; Mohamed Zahran, MD, Principal Investigator — Urology and Nephrology center; Mahmoud Laimon, MSc, Principal Investigator — Urology and Nephrology center; Hossam Nabeeh, Msc, Principal Investigator — Urology and Nephrology center; Mohamed Abdulatif, Msc, Principal Investigator — Urology and Nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Ahmed Shoma, MD, Phd (Study Chair)